CLINICAL TRIAL: NCT07157397
Title: Effect of Plant-Focused Diet on Nutritional Status of Malnourished Patients Undergoing Peritoneal Dialysis in a Selected Hospital Care Setting
Brief Title: Effect of a Plant-Focused Diet on Nutritional Status in Malnourished Peritoneal Dialysis Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Principal Investigator, Harvinder Kaur A/P Gilcharan Singh, Principal Investigator, National University of Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GGPM-2024-051
Record Dates: First submitted 2025-08-14; First posted 2025-09-05 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: End Stage Renal Disease (ESRD); End Stage Kidney Disease (ESRD); Peritoneal Dialysis (PD); Malnourished
Keywords: Peritoneal Dialysis; End Stage Renal Disease; End Stage Kidney Disease; Malnutrition; Plant-Focused Diet; Plant-Based Diet; Nutritonal Status; Dietary Counselling; Quality of Life; Physical Fitness; Inflammation; Appetite; Malaysia; Nutritional Intervention
MeSH Terms: conditions — Kidney Failure, Chronic; Malnutrition; Inflammation

STUDY DESIGN:
Intervention Model Description: Participants are randomly allocated to one of two groups: a plant-focused diet group or a standard-of-care renal diet group. Each participant will remain in their assigned group for the entire 6-month intervention period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-Focused Diet (Experimental): Participants will receive individualised diet counselling and sample meal plans emphasizing plant-based protein sources while meeting recommended protein and energy requirements for peritoneal dialysis patients. Patients in this group will be required to consume plant-focused meals for the majority of their daily meals. For example, those consuming 3 meals per day must ensure that at least 2 out of the 3 meals are plant-based, while those consuming 4 meals per day must ensure that at least 3 out of the 4 meals are plant-based. The remaining meal or snack may include either plant- or animal-based foods to support flexibility and adherence. The diet will be tailored to each patient's nutritional status and dialysis prescription, with monthly follow-ups from a dietitian to monitor adherence and provide adjustments as needed.
  Interventions: Behavioral: Plant-Focused Diet Counselling
- Standard-of-Care Renal Diet (Active Comparator): Participants will receive the current standard-of-care renal diet for peritoneal dialysis patients and be encouraged to maintain their usual dietary and physical activity patterns, with guidance to ensure that at least 50% of their total protein intake comes from high biological value (HBV) animal-based sources. The diet will be tailored to each patient's nutritional status and dialysis prescription, with monthly follow-ups from a dietitian to monitor adherence and provide adjustments as needed.
  Interventions: Behavioral: Standard Renal Diet Counselling

INTERVENTIONS:
Behavioral: Plant-Focused Diet Counselling — Individualized dietary counseling conducted with the use of sample meal plans and infographics to guide patients to consume a diet emphasising plant-based protein sources while meeting nutritional requirements for peritoneal dialysis patients.
  Arms: Plant-Focused Diet
Behavioral: Standard Renal Diet Counselling — Individualized dietary counseling conducted with the use of sample meal plans and infographics based on current guideline recommendations, to guide patients to consume a diet emphasising animal-based protein sources while meeting nutritional requirements for peritoneal dialysis patients.
  Arms: Standard-of-Care Renal Diet

SUMMARY:
The goal of this clinical trial is to determine whether a plant-focused diet improves nutritional and health outcomes of malnourished adults undergoing peritoneal dialysis (PD). It will also learn about the safety of this diet in this population.

The main questions it aims to answer are:

1. Does a plant-focused diet improve nutritional status compared to a standard kidney diet in PD patients?
2. What changes occur in anthropometric, biochemical, and dietary measures over 6 months?

Researchers will compare the plant-focused diet to a standard-of-care renal diet to see which is more effective in improving nutrition in PD patients.

Participants will:

* Be randomly assigned to follow the plant-focused diet or the standard diet.
* Be monitored for 6 months through in-person visits (aligned with their routine clinic appointments) and virtual check-ins via messages or calls.
* Have their progress monitored for changes in outcomes such as nutrition, blood tests, kidney function, and quality of life.

DETAILED DESCRIPTION:
End-stage renal disease (ESRD) is a growing health concern in Malaysia, with a significant increase in the proportion of patients receiving peritoneal dialysis (PD) from 13.0% in 2014 to 18% in 2023. While PD offers certain clinical advantages, it is associated with common complications such as malnutrition and protein-energy wasting (PEW), which contribute to poor patient outcomes.

Emerging evidence suggests that plant-focused diets may have beneficial effects on nutritional status, inflammation, and metabolic complications in PD patients. However, data on their safety, efficacy, and long-term impact in this population remain limited. Hence, this study aims to address this research gap.

This study is a randomized, open-label clinical trial that will compare the effects of a plant-focused diet to a standard-of-care renal diet in malnourished PD patients over a 6-month period.

Participants will be recruited from Hospital Canselor Tuanku Muhriz (HCTM) UKM and randomized into two groups. Both groups will receive individualised dietary counselling and will be followed-up according to their assigned diet plan. Monitoring will occur through physical visits aligned with routine clinic visits, and through virtual check-ins (messages or phone calls). Key outcomes will be measured at baseline, 3 months, and 6 months.

The objectives of this study is:

1. To assess the baseline nutritional status of PD patients in relation to their dietary knowledge, attitude, and practice (KAP), sociodemographic and medical history, anthropometric measurements, biochemical and dietary data, malnutrition-inflammation score (MIS), physical function, quality of life (QOL), and appetite.
2. To compare changes in primary outcomes consisting of dietary adequacy, dialysis adequacy, and kidney function, between groups after 3 and 6 months of intervention.
3. To compare changes in secondary outcomes consisiting of anthropometric measurements, biochemical data, inflammatory markers, adherence to the dietary regime, MIS, physical function, QOL, appetite, and retention rate, between groups after 3 and 6 months.

The findings of this trial may provide important evidence to guide nutritional recommendations for PD patients, improve nutritional outcomes, and address common misconceptions that may contribute to poor dietary intake in this population.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients (>18 years old), attending HTCM PD clinic visits
* Have undergone peritoneal dialysis for at least 6 months
* Have a serum albumin level <40 g/L
* Have a BMI of < 25 kg/m2
* Have a malnutrition inflammation score (MIS) of mild, moderate or severe
* Agreed to follow the dietary instructions based on the randomization assignment
* Agreed to attend baseline visits and additional follow-up appointments at months 1, 3, and 6 post- randomization, either in person or via telehealth, and respond to monthly or more frequent phone calls

Exclusion Criteria:

* Have been hospitalized for the past 3 months
* Have ongoing infection/sepsis
* Has undergone surgery in the past 6 months
* Have high inflammatory diseases, malignancy, or cancer
* Have dialysis adequacy of <1.2 Kt/V

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-01-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in Dietary Adequacy | At baseline, after 3 months of intervention, and after 6 months of intervention
  Dietary intake collected from analysis of 3-day dietary recalls (2 weekdays, 1 weekend), using Nutritionist Pro software.
  Dietary adequacy is assessed based on the comparison of each participant's macro- and micro-nutrient intakes against their estimated nutrient requirements. A deviation of more than 20% from the requirement will be classified as dietary inadequacy. Data will be summarised as percentage of participants meeting vs. not meeting adequacy.
Changes in Dialysis Adequacy | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Dialysis adequacy will be assessed using weekly Kt/V (urea), obtained from patients' medical records. A total Kt/V < 1.7 will be considered indicative of inadequate dialysis.
Changes in Concentration of Urea | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Concentration of Creatinine | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in µmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Concentration of Sodium | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Concentration of Potassium | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Concentration of Phosphate | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Concentration of Serum Albumin | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in g/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Concentration of Total Protein | At baseline, after 3 months of intervention, and after 6 months of intervention.
  A renal function parameter, measured in g/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.

SECONDARY OUTCOMES:
Changes in Weight | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Post-dialysis weight will be measured in kilograms (kg), using a digital scale, with patients wearing light clothing and no heavy objects.
Height | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Height will be measured in centimeters (cm), with patients standing straight on the stadiometer, following the Frankfurt horizontal plane.
Changes in Body mass index (BMI) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Body mass index will be calculated by dividing weight (kg) by the square of height (m²), recorded as kg/m².
Changes in Triceps skinfold (TSF) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Triceps skinfold will be assessed using skinfold callipers, recorded in centimetres (cm).
Changes in Dietary Adherence/Compliance | Baseline and monthly, for up to 6 months.
  Patients will be required to complete a 3-day food diary (2 weekdays and 1 weekend). Food diaries will be reviewed monthly, either in person at clinic visits or remotely via phone or messaging, and will be scored using the binary dietary compliance scoring system developed specifically for this study. Using the scoring system (maximum score = 21), a total score of <10.5 out of 21 (<50%) will be classified as poor compliance, while a score of ≥10.5 out of 21 (≥50%) will be considered adequate. Scores range from 0 - 21, with higher scores indicating better compliance.
  The scoring system will be pilot tested with patients during the first 2 weeks of the study period.
Changes in Malnutrition-Inflammation Score (MIS) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Each component (medical history, physical examination, BMI, and laboratory markers) is scored from 0 (normal nutrition status) to 3 (severe nutritional deficit). Total scores range from 0 to 30, with higher scores indicating higher degrees of malnutrition. A score of <5 indicates normal nutritional status, while ≥5 signifies malnutrition.
Changes in Appetite and Food Satisfaction (AFSQ) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Evaluated using the Appetite and Food Satisfaction Questionnaire (AFSQ). Consists a facial hedonic scale to assess appetite levels and five additional questions. Each question is scored from 0 to 3, with a total score ranging from 0 to 18 and lower scores indicate better appetite and food satisfaction.
Changes in Quality of life (WHOQOL-BREF) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Evaluated using the World Health Organization Quality of Life-BREF (WHOQOL-BREF). It consists of 26 items categorized into four domains: physical health, psychological well-being, social relationships, and environment. Each item is rated on a 5-point Likert scale, and domain scores are calculated as the mean of their respective items. Raw domain scores are transformed to a 4-20 scale and further converted to a 0-100 scale to facilitate interpretation, with higher scores indicating better QOL
Changes in Physical Function (SPPB) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Assessed using the Short Physical Performance Battery (SPPB), with scores calculated and higher total scores indicating better physical function. Muscular strength will be measured using the Jamar handgrip dynamometer.
Changes in Physical Activity Levels (IPAQ-SF) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Evaluated using the International Physical Activity Short Form questionnaire. Total scores are calculated by summing the duration and frequency of all activities, while domain-specific and activity-specific sub scores are also determined. The collected data will be reported as either a continuous measure or in metabolic equivalents (METs) per minute.
Retention Rate | End of study (after 6 months of intervention).
  The retention rate will be calculated as the percentage of participants who complete the 6-month study period. The number of participants completing the study will be divided by the total number enrolled and multiplied by 100.
Mid-upper arm circumference (MUAC) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Mid-upper arm circumference will be measured using a measuring tape, recorded in centimetres (cm).
Mid-arm muscle circumference (MAMC) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Mid-arm muscle circumference (MAMC) will be calculated using the formula: MAMC = MUAC - (π × TSF). Measurements will be recorded in centimetres (cm). It serves as an anthropometric indicator of muscle mass and is used as a proxy for lean body mass when bioelectrical impedance analysis (BIA) is unavailable. A lower MAMC reflects reduced muscle reserves and potential malnutrition.
Changes in Total cholesterol | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Serum total cholesterol, a parameter of the lipid profile, will be recorded in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges
Changes in Triglycerides | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Serum tryglycerides, a parameter of the lipid profile, will be recorded in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges
Changes in High-density lipoprotein cholesterol (HDL-C) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Serum High-density lipoprotein cholesterol (HDL-C), a parameter of the lipid profile, will be recorded in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges
Changes in Low-density lipoprotein cholesterol (LDL-C) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Serum Low-density lipoprotein cholesterol (LDL-C), a parameter of the lipid profile, will be recorded in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges
Changes in Glycated haemoglobin (HbA1c) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Glycated haemoglobin (HbA1c), a parameter of the blood glucose profile, will be recorded in %, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Fasting Blood Glucose (FBG) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Fasting Blood Glucose (FBG), a parameter of the blood glucose profile, will be recorded in mmol/L, obtained from medical records. Results will be compared against standard laboratory reference ranges.
Changes in Serum Total Iron Binding Capacity (TIBC) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Serum Total Iron Binding Capacity (TIBC), an inflammatory marker, will be obtained from medical records and recorded in µmol/L. Results will be compared against standard laboratory reference ranges.
Changes in Serum High-sensitivity C-reactive protein (hsCRP) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Serum hsCRP, an inflammatory marker, will be measured in mg/L. A 10 mL fasting blood sample (following a 12-hour overnight fast) will be collected by trained hospital staff using automated procedures. Samples will be analysed at an external accredited laboratory (Innoquest). Results will be compared against standard laboratory reference ranges.
Changes in Normalised protein catabolic rate (nPCR) | At baseline, after 3 months of intervention, and after 6 months of intervention.
  Normalised protein catabolic rate (nPCR), a protein intake indicator, will be obtained from medical records and recorded in g/kg/day. Results will be compared against standard laboratory reference ranges.
Dietary Knowledge, Attitude, and Practice (KAP) Questionnaire | At baseline.
  Participants will complete a 34-item questionnaire adapted from a validated tool used in haemodialysis patients. It includes three subscales: knowledge (12 items), attitude (7 items), and practice (15 items). Knowledge items are scored 0-1 (correct/incorrect), while attitude and practice items are rated on a 0-4 Likert scale. Total scores range from 0 to 100, with higher total scores indicating better dietary KAP.
Changes in body fat percentage (%) | At baseline, 3 months, and 6 months.
  Body fat percentage will be measured in percentage (%) using a bioelectrical impedance analysis (BIA) device.
Changes in Fat-free mass (kg) | At baseline, 3 months, and 6 months.
  Fat-free mass will be assessed using a bioelectrical impedance analysis (BIA) device, recorded in kilograms (kg).
Changes in skeletal muscle mass (kg) | At baseline, 3 months, and 6 months.
  Skeletal muscle mass will be measured using a bioelectrical impedance analysis (BIA) device, recorded in kilograms (kg).
Changes in fat mass (kg) | At baseline, 3 months, and 6 months.
  Fat mass will be measured using a bioelectrical impedance analysis (BIA) device, recorded in kilograms (kg).

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Canselor Tuanku Muhriz UKM, Cheras, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to confidentiality requirements and to protect participant privacy. Only aggregated, de-identified results will be published.